CLINICAL TRIAL: NCT01699880
Title: High Flow Nasal Cannula Oxygen for Pre and During Procedure Oxygenation During Tracheal Intubation: Comparison With High FiO2 Non Rebreathing Bag Reservoir Facemasks
Brief Title: Efficacy of High Flow Nasal Cannula Oxygen to Reduce Desaturation During Tracheal Intubation
Acronym: HAPI
Status: Completed | Type: Observational
Sponsor: Hôpital Louis Mourier (Other)
Responsible Party: Principal Investigator, Prof Jean-Damien RICARD, Professor of Intensive Care Medicine, assistant head of ICU, Hôpital Louis Mourier
Other Study IDs: HLM_JDR1
Record Dates: First submitted 2012-10-01; First posted 2012-10-04 (Estimated); Last update posted 2014-08-12 (Estimated); Status verified 2014-08

CONDITIONS: Need for Intubation; Oxygenation Before and During Intubation
Keywords: tracheal intubation; preoxygenation; desaturation; hypoxemia; oxygen therapy; high flow nasal cannula oxygen therapy
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- conventional high FiO2 bag reservoir facemask: this group of patients is intubated according to our current practice that requires the use of a high FiO2 nonrebreathing with bag reservoir facemask to ensure preoxygenation in patients requiring tracheal intubation. a small nasal catheter is inserted just before laryngoscopy to ensure a low oxygen flow to allow oxygenation during laryngoscopy.
- high flow nasal cannula oxygen: we wish to change our standard practice of preoxygenation and expand our use of high flow nasal cannula oxygen therapy to the tracheal intubation setting. Currently, used of high flow oxygen nasal cannula oxygen therapy to ensure oxygenation during intubation is limited to the patients already under high flow nasal cannula oxygen. the change of practice consists in the systematic use of high flow nasal cannula oxygen therapy in all patients requiring tracheal intubation in the ICU.

SUMMARY:
Tracheal intubation of critically ill patients is associated in the intensive care unit (ICU) with significant complications and morbidity. Patient desaturation is one of the most common complications that may lead to cardiac arrest despite pre-intubation oxygenation. Preoxygenation can be improved by the use of non-invasive ventilation, but this technique can be cumbersome to implement in the context of urgent intubation and more importantly it does not insure oxygenation during intubation. High flow nasal cannula oxygen therapy is a technique that has been shown to improve patient oxygenation in the context of acute hypoxemic respiratory failure. It bears the potential to be of clinical benefit in the setting of tracheal intubation in the ICU to ensure patient safety. The purpose of this study is to compare pre- and per-intubation (during intubation) oxygenation with either a conventional high FiO2 oxygen bag reservoir facemask (current standard practice) or high flow nasal cannula oxygen therapy (new practice to be implemented in our ICU).

DETAILED DESCRIPTION:
Pre-oxygenation is ensured in our ICU with a high FiO2 nonrebreathing facemask, except in patients already under high flow nasal cannula oxygen therapy because of acute hypoxemic respiratory failure. A nasal catheter is positioned to ensure a low oxygen flow during laryngoscopy. Whether or not all patients should benefit from high flow nasal cannula oxygen therapy for pre-oxygenation remains unknown. In order to improve quality of care delivered to our patients and in anticipation of a change in our practice, we decided to record prospectively oxygen parameters during and immediately of intubation using a facemask and to compare them with parameters obtained in patients intubated after our change in practice. The change of practice consists in the systematic use of high flow nasal cannula oxygen therapy to ensure pre and during procedure (tracheal intubation)oxygenation.

ELIGIBILITY:
Inclusion Criteria:

* ICU patient requiring tracheal intubation

Exclusion Criteria:

* age < 18 years
* cardiac arrest
* acute respiratory failure requiring immediate high flow nasal cannula oxygen, defined as patient with SpO2 < 95% while under 15 L:min oxygen with a nonrebreathing facemask

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU patients requiring tracheal intubation
Sampling Method: Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2011-03; Primary Completion 2012-11 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
lowest pulse oxymetry (SpO2) during intubation | from beginning of laryngoscopy to completed intubation
mean pulse oxymetry during intubation | from beginning of laryngoscopy to completed intubation
pulse oxymetry after preoxygenation | 3min prexoxygenation
pulse oxymetry after intubation | at connection of the patient to the ventilator

SECONDARY OUTCOMES:
mean pulse oxymetry | one, five and thirty minutes after intubation
number of pulse oxymetry below 90% | from laryngoscopy to 30 minutes once tracheal intubation completed
number of pulse oxymetry below 80% | from laryngoscopy to 30 minutes once tracheal intubation completed

OTHER OUTCOMES:
cardiac arrest | during and immediately after procedure
hemodynamic instability defined as arterial systolic blood pressure below 80 mmHg | during and immediately after procedure

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Damien Ricard, MD, PhD, Principal Investigator — Hopital Louis Mourier, AP-HP, Colombes, France
Locations (1):
- Medico-surgical ICU, Colombes, France

REFERENCES:
- [Background] Sztrymf B, Messika J, Bertrand F, Hurel D, Leon R, Dreyfuss D, Ricard JD. Beneficial effects of humidified high flow nasal oxygen in critical care patients: a prospective pilot study. Intensive Care Med. 2011 Nov;37(11):1780-6. doi: 10.1007/s00134-011-2354-6. Epub 2011 Sep 27. PMID 21946925
- [Background] Ricard JD. High flow nasal oxygen in acute respiratory failure. Minerva Anestesiol. 2012 Jul;78(7):836-41. Epub 2012 Apr 24. PMID 22531566
- [Background] Sztrymf B, Messika J, Mayot T, Lenglet H, Dreyfuss D, Ricard JD. Impact of high-flow nasal cannula oxygen therapy on intensive care unit patients with acute respiratory failure: a prospective observational study. J Crit Care. 2012 Jun;27(3):324.e9-13. doi: 10.1016/j.jcrc.2011.07.075. Epub 2011 Sep 29. PMID 21958974
- [Background] Lenglet H, Sztrymf B, Leroy C, Brun P, Dreyfuss D, Ricard JD. Humidified high flow nasal oxygen during respiratory failure in the emergency department: feasibility and efficacy. Respir Care. 2012 Nov;57(11):1873-8. doi: 10.4187/respcare.01575. Epub 2012 Mar 13. PMID 22417844
- [Derived] Miguel-Montanes R, Hajage D, Messika J, Bertrand F, Gaudry S, Rafat C, Labbe V, Dufour N, Jean-Baptiste S, Bedet A, Dreyfuss D, Ricard JD. Use of high-flow nasal cannula oxygen therapy to prevent desaturation during tracheal intubation of intensive care patients with mild-to-moderate hypoxemia. Crit Care Med. 2015 Mar;43(3):574-83. doi: 10.1097/CCM.0000000000000743. PMID 25479117